CLINICAL TRIAL: NCT01172613
Title: Optimal Concentration of Allergen Extract of Dermatophagoides Pteronyssinus to be Used in Diagnostic Allergy Skin Prick Test Among Thai Population
Brief Title: Optimal Concentration of Dermatophagoides Pteronyssinus (Dp) Allergen Extract for Skin Prick Test (SPT) of Thai Population
Acronym: DSPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Professor Pakit Vichyanond, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Other Study IDs: 112/2553(EC3)
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Skin Prick Test
Keywords: allergic rhinitis; concentration of diagnostic reagent; allergen extract, house dust mites (Dp); skin prick test; nasal allergen provocation test
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy subjects no symptoms
- allergic rhinitis patient

SUMMARY:
The purpose of this study is to determine the appropriate concentration of diagnostic reagent of house dust mite (Dp) to be used in diagnostic allergy skin prick test among Thai population with allergic rhinitis.

DETAILED DESCRIPTION:
The current allergy diagnostic reagent of house dust mites marketed in the USA is at 10,000 AU/ml. This is based on the IDEAL50 concept put forth by Turkeltaub et al, almost 3 decades ago. Such concentration has been shown to give large degree of false positives even in the US population.

In Thailand, it was anecdotally observed that at such concentration, sizes of positive tests among atopic subjects were quite large and could lead to discomfort and a possible anaphylaxis in certain allergic individuals. Moreover, up to 40% of normal individuals could give positive reaction to this concentration.

It is therefore desirable to reexamine the appropriate concentration of diagnostic reagent of house dust mites among the Thai population and will be the main objective of this research.

ELIGIBILITY:
Inclusion Criteria:allergic rhinitis

* clinical diagnosis of allergic rhinitis
* has skin prick test positive to standard Dp extract (wheal diameter 3 mm. or greater)
* not take any medications that interfere the tests (skin prick test and nasal allergen provocation test)

Inclusion Criteria:healthy subject

* no underlying disease
* not take any medications that interfere the tests (skin prick test and nasal allergen provocation test)

Exclusion Criteria:

* has skin prick test positive to standard Dp extract with wheal diameter more than 10 mm.
* has chronic disease eg. HIV infection, neurological diseases, hypertension, cardiac diseases, pulmonary diseases, hepatobiliary diseases, renal diseases, endocrinological diseases, congenital malformation, malignancy
* if has asthma, uncontrolled asthma symptom or PEF < 70%
* during pregnancy or lactation
* has chronic skin disease
* participate other project within 30 days
* has abnormal anatomy of the nose

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: allergic rhinitis patients in Siriraj hospital (tertiary care) control group: healthy subjects from community sample
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
appropriate concentration of diagnostic reagent of house dust mite (Dp) | 15 minutes
  to determine appropriate dilutional concentration of diagnostic reagent of house dust mite (Dp) that has high sensitivity and positive predictive value and wheal size not more than 10 mm. to be used in diagnosis allergic rhinitis in Thai population by skin prick test.

SECONDARY OUTCOMES:
false positive rates of various dilutions of diagnostic reagent (house dust mite: Dp) that be used in skin prick test in Thai healthy population | 15 minutes
false negative rates of various dilutions of diagnostic reagent (house dust mite: Dp) that be used for diagnosis allergic rhinitis in Thai population by skin prick test | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Professor Pakit Vichyanond, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand